CLINICAL TRIAL: NCT05234866
Title: Paradoxical Lucidity in Severe End-Stage Dementia
Status: Recruiting | Type: Observational
Sponsor: NYU Langone Health (Other)
Collaborators: National Institute on Aging (NIA) (NIH)
Responsible Party: Sponsor
Other Study IDs: 20-01854
Record Dates: First submitted 2022-01-31; First posted 2022-02-10 (Actual); Last update posted 2025-08-14 (Actual); Status verified 2025-08

CONDITIONS: Dementia
MeSH Terms: conditions — Dementia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Phase I (Feasibility Study)
- Phase II (Prospective Study)

SUMMARY:
Cognitive decline in dementia is considered irreversible, however episodes of paradoxical lucidity (PL) in severe dementia suggest other mechanisms may be in play. Beyond anecdotal reports of transient PL events occurring in patients predominantly in late-stage dementia and typically lasting anywhere from a few minutes to several hours, little is known about PL. The study team proposes to develop and conduct a mixed methods prospective study of PL during end stage advanced dementia, creating a definition and measurement scale for PL in advanced dementia, and identifying the potential electro cortical biomarkers of PL in advanced dementia. This study will be divided in two phases: Phase I and Phase II. During Phase I, the study team will collect sufficient and necessary data through an online survey and focus groups as well as assess the safety and feasibility of using symptom diaries (also known as daily trackers or journals) and real-time video EEG monitoring (vEEG). After preliminary review of the study procedures, the PI will decide whether to move onto the Phase II. The second phase will aim to expand the study population and refine study methods as well as create a definition and measurement scale for PL in advances dementia.

ELIGIBILITY:
Inclusion Criteria:

* Age > 18 years
* Advanced (severe) dementia diagnosed using the Global Deterioration Scale (GDS) with a score of 7 or the Palliative Performance Scale (PPS) with a score of less than 30%
* Accepted for hospice care based on the Medicare eligibility guidelines
* No longer being provided with nutrition or fluids
* Anuria (dry diaper) or less than 200cc urine (almost dry diaper) in any 24-hour period

Exclusion Criteria:

* Cognitive or functional impairment due to a diagnosis other than dementia
* Dementia with a GDS score <7 (mild, moderate, moderately severe dementia). Please refer to rationale outlined for inclusion criteria 2.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: 1. Adults over 18 years of age diagnosed with advanced dementia
  2. Hospice workers, geriatric, palliative care physicians and other healthcare providers
  3. Family, friends and caregivers
Sampling Method: Non-Probability Sample
Enrollment: 520 (Estimated)
Dates: Start 2022-06-02 (Actual); Primary Completion 2026-03-31 (Estimated); Study Completion 2026-05-31 (Estimated)

PRIMARY OUTCOMES:
Phase I and II - Number of self-reports of patient distress/discomfort in relation to symptom diary use and recording of potential episodes of paradoxical lucidity (PL) using mobile devices | up to Day 7
Phase I - Number of self-reports of informants' distress or discomfort due to the presence of the video EEG device. | up to Day 7
Phase I - Number of families who express interest in the study and contact the research team | up to Day 7
Phase I - Number of successful informed consents obtained from family members/legally authorized health care proxies | up to Day 7
Phase I - Number of days taken for patients to die after being identified by hospice staff with a life expectancy </= 7 days | up to Day 7
Phase I - Number of diary reports completed and returned to research staff | up to Day 7
Phase I - Time taken to establish video EEG monitoring in homes or nursing homes | up to Day 7
Phase I - Total number of instances in which video EEG monitoring was successfully initiated | up to Day 7
Phase I - Average number of days for which video EEG monitoring was completed | up to Day 7

SECONDARY OUTCOMES:
Phase II - Change in average number of changes in EEG rhythm | Baseline, up to Day 7
Phase II - Average number of changes in EEG rhythm during PL | Baseline, up to Day 7

CONTACTS AND LOCATIONS:
Overall Officials: Sam Parnia, MD, PhD, Principal Investigator — NYU Langone Health
Locations (1):
- NYU Langone Health, New York, New York, United States

IPD SHARING:
Plan to Share IPD: Yes
Individual participant data that underlie the results reported in this article, after deidentification (text, tables, figures, and appendices) will be shared upon reasonable request.
Supporting Information: Study Protocol, SAP
Time Frame: Beginning 9 months and ending 36 months following article publication or as required by a condition of awards and agreements supporting the research.
Access Criteria: The investigator who proposed to use the data will have access to the data upon reasonable request. Requests should be directed to Sam.Parnia@nyulangone.org. To gain access, data requestors will need to sign a date access agreement.